CLINICAL TRIAL: NCT02155348
Title: Comparison Between Bilateral Multifocal Intraocular Lenses and Pseudophakic Monovision: a Randomised Controlled Trial
Brief Title: Comparison Between Bilateral Multifocal Intraocular Lenses and Pseudophakic Monovision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prim. Prof. Dr. Oliver Findl, MBA, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lentis
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multifocal group (Active Comparator): Bilateral cataract surgery with implantation of multifocal IOLs
  Interventions: Procedure: Bilateral cataract surgery with implantation of multifocal IOLs; Device: Lentis LS-313
- Monovision (Active Comparator): Bilateral cataract surgery with monovision
  Interventions: Procedure: Bilateral cataract surgery with monovision; Device: Lentis LS-313

INTERVENTIONS:
Procedure: Bilateral cataract surgery with implantation of multifocal IOLs — Lentis LS-313, multifocal, target refraction of the distance-dominant eye: 0.00D, target refraction of the other eye: -0.50D
  Arms: Multifocal group
Procedure: Bilateral cataract surgery with monovision — Lentis L-313, monofocal, target refraction of the distance-dominant eye: 0.00D to -0.25D, target refraction of the other eye: -1.50D
  Arms: Monovision
Device: Lentis LS-313

SUMMARY:
More and more patients like to achieve complete spectacle independence after cataract surgery. Two possibilities that are particularly often used today are on the one hand multifocal lenses, and on the other hand the concept of monovision (in doing so one eye is adjusted for closeness and the other focuses for distance). The drawback with multifocal lenses is that some patients are bothered by glare phenomena, the disadvantage of monovision is that some patients lose a little of their stereo vision.

The aim of this study is a direct comparison of these two methods. Therefore 70 patients are included in 2 groups. In one group, patients receive on both sides a multifocal IOL with a near addition of +1.5 D and the patients in the second group receive monovision. One hour, 1 week and 3 months after surgery, patients are invited and tests for visual accuity are performed for near vision (40cm), intermediate vision (80cm) and distant vision (400cm). Furthermore, contrast sensitivity and stereopsis of patients is assesed. Additional measurements for detecting the tilt of the lens will be performed.

DETAILED DESCRIPTION:
Spectacle independence is a central aim in modern cataract surgery. Although bilateral monofocal IOL implantation, aiming for emmetropia or low myopia, leads to high levels of patient satisfaction in distance vision, spectacle dependence for reading and other near vision tasks is the usual result.

The current technique available to surgeons to reduce spectacle dependence is to use bilateral multifocal IOLs. However, a variable number of patients do complain of problems with glare, haloes and lights especially in the hours of darkness (dysphotopsia symptoms). Dysphotopsia symptoms may vary significantly from patient to patient. The real incidence of dysphotopsia like symptoms after cataract surgery and multifocal IOL is unknown 6 and the implantation of multifocal IOLs is a commonly accepted contraindication in patients who are night drivers.

Another option to allow spectacle independence is monovision. Monovision is where one eye can see clearly in the distance and the other eye is intentionally made short-sighted so that it has either near reading vision (full monovision) or intermediate (arms length) or distance vision (limited monovision). Monovision has two major advantages, very little dysphotopsia and it is cheaper compared to multifocal IOLs. However, disadvantages are a reduced stereopsis and there is a need for neuroadaptation.

The rationale of this trial was to compare bilateral multifocal intraocular lenses (MIOLs) with monovision after cataract surgery concerning visual function and spectacle independence.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract
* Scheduled for bilateral cataract extraction
* Motivated to be less spectacle dependant
* Age 21 and older
* Corneal astigmatism ≤ 1.5 D (Keratometry, IOL Master 500)
* written informed consent prior to recruitment

Exclusion Criteria:

* Pregnancy (pregnancy test will be taken pre-operatively in women of reproductive age)
* Retinitis pigmentosa
* Chronic uveitis
* Amblyopia
* Pupil decentration > 1mm center shift
* preceded retinal surgery
* preceded Laser-in-situ-Keratomileusis (LASIK)
* Any ophthalmic abnormality that could compromise visual function or the measurements

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-01 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Spectacle independence of patients with bilateral multifocal intraocular lenses in comparison to patients with pseudophakic monovision evaluated using a questionnaire | 3 months

SECONDARY OUTCOMES:
Uncorrected and Best Corrected Distance Visual Acuity, Uncorrected and Distance Corrected Intermediate Visual Acuity, Uncorrected and Distance Corrected Near Visual Acuity between the test and the control group | 3 months
Reading Speed | 3 months
Stereo Vision and Contrast Sensibility | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- VIROS - Vienna Institute for Research in Ocular Surgers - Departement of Opthalmology - Hanusch Hospital, Vienna, Vienna, Austria